CLINICAL TRIAL: NCT04157933
Title: A Placebo-Controlled, Double-Blind, Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Profile of AZ-009 in Subjects With Established Parkinson's Disease
Brief Title: Staccato Apomorphine Multi-dose PK and PD in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-009-102
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2019-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Crossing Over, Genetic

STUDY DESIGN:
Intervention Model Description: This study will be conducted in subjects with established Parkinson's disease in 2 parts. Part A will examine the tolerability, safety, and pharmacokinetics of AZ-009 dose escalation ; and Part B will assess the tolerability, safety, pharmacokinetics, and pharmacodynamics of AZ-009 compared with placebo in a crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- A-1a (Experimental): Part A, Arm 1 (active), Dose 1 (009-A1)
  Interventions: Drug: 009-A1
- A-2a (Experimental): Part A, Arm 2 (active), Dose 2 (009-A2)
  Interventions: Drug: 009-A2
- A-3a (Experimental): Part A, Arm 3 (active), Dose 3 (009-A3)
  Interventions: Drug: 009-A3
- A-0p (Placebo Comparator): Part A, placebo comparator in all 3 arms, placebo dose (009-A0)
  Interventions: Drug: 009-A0
- B-1 (009-B3 -> 009-B0) (Experimental): Crossover (active to placebo)
  Interventions: Drug: 009-B1 (active --> placebo) crossover
- B-1 (009-B0 -> 009-B3) (Experimental): Crossover (placebo to active)
  Interventions: Drug: 009-B2 (placebo --> active) crossover

INTERVENTIONS:
Drug: 009-A1 — Inhaled apomorphine via Staccato aerosol, Dose 1 (low dose) each day for first 5 days, then 3 doses Dose 1 (low dose) q 2 hr on Day 6
  Arms: A-1a
Drug: 009-A2 — Inhaled apomorphine via Staccato aerosol, Dose 2 (middle dose) each day for first 5 days, then 3 doses Dose 2 (middle dose) q 2 hr on Day 6
  Arms: A-2a
Drug: 009-A3 — Inhaled apomorphine via Staccato aerosol, Dose 3 (high dose) each day for first 5 days, then 3 doses Dose 3 (high dose) q 2 hr on Day 6
  Arms: A-3a
Drug: 009-A0 — Inhaled placebo via Staccato aerosol, Dose 0 (placebo) each day for first 5 days, then 3 doses Dose 0 (placebo) q 2 hr on Day 6
  Arms: A-0p
Drug: 009-B1 (active --> placebo) crossover — Up to 2 doses (Dose 3) ; minimum of 2 hrs between doses, on Day 1, followed by Up to 2 doses (placebo) ; minimum of 2 hrs between doses, on Day 2
  Arms: B-1 (009-B3 -> 009-B0)
Drug: 009-B2 (placebo --> active) crossover — Up to 2 doses (placebo) ; minimum of 2 hrs between doses, on Day 1, followed by Up to 2 doses (Dose 3) ; minimum of 2 hrs between doses, on Day 2
  Arms: B-1 (009-B0 -> 009-B3)

SUMMARY:
This study will be conducted in subjects with established Parkinson's disease in 2 parts. Part A will examine the tolerability, safety, and pharmacokinetics of AZ-009 dose escalation ; and Part B will assess the tolerability, safety, pharmacokinetics, and pharmacodynamics of AZ-009 compared with placebo in a crossover design

DETAILED DESCRIPTION:
This study will be conducted in subjects with established Parkinson's disease in 2 parts.

Part A will examine the tolerability, safety, and pharmacokinetics of daily doses of AZ-009 for 5 days followed by 3 doses on each of days 6 and 7 in dose escalation through 3 cohorts

Part B will assess the tolerability, safety, pharmacokinetics, and pharmacodynamics of AZ-009 compared with placebo in subjects with established Parkinson's disease experiencing regular OFF episodes

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 30 and 85 years of age, inclusive at the time of signing the informed consent document with a clinical diagnosis of Parkinson's Disease
* Body weight ≥ 50 kg and BMI within the range of 18 to 32 kg/m2.
* Willing and able to be confined at the clinical research center for the study period and adhere to overall study visit schedule, procedures and other protocol requirements.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

* Any significant medical condition, psychiatric illness or history of depression that could, in the investigator's opinion, compromise the subject's safety or interfere with the completion of this protocol.
* History of clinically significant central nervous system, cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions including gastric bypass or other weight loss

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
A - Dose Proportionality of multi-dose inhaled apomorphine by Power Analysis of AUC | 6 days
  Dose proportionality of inhaled Staccato apomorphine AUC across all 3 doses during Days 1-5 and multiple daily dosing (all 3 doses q 2 hr per day) on Day 6 using a power model [regression of log(AUC) versus log(dose)] in subjects with established Parkinson's disease
B1 - Effect on MDS-UPDRS in Parkinson's disease OFF periods | 2 days
  Explore in a crossover design on consecutive days the pharmacodynamics of AZ-009 compared with placebo on the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III in subjects with established Parkinson's disease experiencing regular OFF episodes.
B2 - Effect on Physician Disease State Assessment in Parkinson's disease OFF periods | 2 days
  Explore in a crossover design on consecutive days the pharmacodynamics of AZ-009 compared with placebo on the Physician Disease State Assessment in subjects with established Parkinson's disease experiencing regular OFF episodes.
B3 - Effect on Patient Assessment of ON/OFF in Parkinson's disease OFF periods | 2 days
  Explore in a crossover design on consecutive days the pharmacodynamics of AZ-009 compared with placebo on Patient Assessment of ON/OFF in subjects with established Parkinson's disease experiencing regular OFF episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Geert J Groeneveld, MD, PhD, Principal Investigator — Center for Human Drug Research (The Netherlands)
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands